CLINICAL TRIAL: NCT02531386
Title: System Accuracy Evaluation of Accu-Chek Aviva Nano (Roche Diagnostics), Accu-Chek Performa Nano (Roche Diagnostics), FreeStyle Lite (Abbott Diabetes Care), OneTouch Verio IQ (LifeScan), Contour Next Link 2.4 (Bayer Consumer Care), One Additional CE-marked Blood Glucose Monitoring System Following ISO 15197:2013
Brief Title: System Accuracy Evaluation of 6 CE-marked Blood Glucose Monitoring System Following ISO 15197:2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1525-BL
Record Dates: First submitted 2015-08-07; First posted 2015-08-24 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

INTERVENTIONS:
Device: 6 blood glucose monitoring systems for self-testing (blood glucose meters)
  Other Names: Accu-Chek Aviva Nano, Accu-Chek Performa Nano, FreeStyle Lite, OneTouch Verio IQ, Contour Next Link 2.4, Accu-Chek Mobile

SUMMARY:
The objective of this study is the evaluation of system accuracy following ISO 15197:2013 (E), clause 6.3 in which accuracy requirements and applicable test procedures for blood glucose monitoring systems intended for self-monitoring of blood glucose by patients are stipulated. In this study, system accuracy evaluation will be performed with CE-marked BGMS (BGMS = Blood Glucose Monitoring System) common among insulin pump users - Accu-Chek Aviva Nano and Accu-Chek Performa Nano (Roche Diagnostics), FreeStyle Lite (Abbott Diabetes Care), OneTouch Verio IQ (LifeScan) Contour Next Link 2.4 (Bayer Healthcare Diabetes Care) and Accu-Chek Mobile with three different reagent system lots for each BGMS.

The study will be performed in 2 parts. Each part will comprise testing of 3 BGMS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or no diabetes
* For provoked blood glucose excursions due to insulin dose adjustment:

  * Male or female with type 1 diabetes or
  * Type 2 diabetes and intensified insulin therapy or insulin pump therapy.
* Minimum age of 18 years
* Signed informed consent form
* Legally competent and capable to understand character, meaning and consequences of the study

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Physical or mental constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Incapability of giving informed consent
* < 18 years
* Legally incompetent
* Accommodated in an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent from investigator or sponsor
* For provoked blood glucose excursions 50 - 80 mg/dl (concentration category 2):
* Coronary heart disease
* Condition after myocardial infarction
* Cerebral incidence
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
System accuracy criteria (see description) | For each subject, the experimental phase has an expected duration of up to 6 hours
  System accuracy criteria
  Following ISO 15197:2013 (E), the BGMS shall meet both of the following criteria:
  Criterion A: 95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 100 mg/dl (5.55 mmol/l) or within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).
  Each lot shall pass acceptability criterion A.
  Criterion B: 99 % of individual glucose measured values shall fall within zones A and B of the Consensus Error Grid (CEG) for type 1 diabetes.
  Applying ISO 15197:2003 accuracy criteria:
  95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 75 mg/dl (4.2 mmol/l) or within ± 20 % at glucose concentrations ≥ 75 mg/dl (4.2 mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany